CLINICAL TRIAL: NCT03239639
Title: A Randomized Control Trial of an Advance Care Planning Intervention to Engaged Substitute Decision-makers in Primary Care
Brief Title: Randomized Control Trial of Advance Care Planning in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Queen's University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 3714
Record Dates: First submitted 2017-08-02; First posted 2017-08-04 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2019-01

CONDITIONS: Chronic Illness
Keywords: Substitute decision makers of patient
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Intervention Model Description: Participants are assigned in 1:1 ratio to intervention or wait list control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Advance care planning education session (Experimental): Delivery of an advance care planning education session at the family doctor's office
  Interventions: Behavioral: Advance care planning education session
- Wait list control (Sham Comparator): The intervention is not provided.
  Interventions: Other: Wait list control

INTERVENTIONS:
Behavioral: Advance care planning education session — Administration of values clarification tool, elicitation of preference for treatment options, if preference for resuscitation, shown an educational video about cardiopulmonary resuscitation, summary document of values and preferences created by a facilitator to share with doctor
  Arms: Advance care planning education session
Other: Wait list control — No intervention
  Arms: Wait list control

SUMMARY:
Sometimes people with health conditions become ill suddenly and can no longer speak for themselves and another person (such as a family member) will make health care decisions for them. This means it is important to think about your wishes and tell others about them. This is called advance care planning. When people have done advance care planning, if they become very sick and cannot speak for themselves they are more likely to get the kind of health care they want and it is easier for the people who make decisions for them. There are tools such as brochures, questionnaires, and videos that can help people learn about these things. This research is being to done to study whether using tools for advance care planning and goals of care discussions will improve how patients and their substitute decision makers do advance care planning. This study is a randomized trial. This means half of the people in this study will meet with someone at their family practice to talk about advance care planning and review some tools and half will get usual care (a Speak Up workbook). The study will 1) evaluate if reviewing the tools, and having help to complete them, helps patients and their substitute decision maker do advance care planning 2) if this intervention will encourage patients to talk to their family doctor about these issues.

DETAILED DESCRIPTION:
In prospective and randomized trials, advance care planning (ACP) significantly improves outcomes including increased likelihood that clinicians and families understand and comply with a patient's wishes, reduces hospitalization at the end of life, results in less intensive treatments at the end of life (according to patients' wishes) and increases use of hospice services. Trials have not been done in primary care. In this project, we aim to determine the efficacy of a care pathway designed to increase the quality and quantity of ACP in patients and their substitute decision-makers in primary care. The study is a multi-site, patient-based, unblinded, randomized trial conducted in family practices in Canada. Participants will be patients who are determined by their physician to be able to benefit from ACP, and the patient's substitute decision-maker. Participant pairs will be randomized to immediate intervention (care pathway) or delayed (8-12 weeks). The intervention is guided use of tools and decision aids to clarify values and preferences for treatments in the event of serious illness or near end of life. The outcomes will be substitute decision-maker engagement in ACP (including self-efficacy for enacting the role), patient engagement in ACP, and decisional conflict.

ELIGIBILITY:
Inclusion Criteria:

* Patients being treated for serious illness in outpatient settings or;
* Patients who could benefit from advance care planning self-assessed or assessed by their physician
* Patient able and willing to identify a substitute decision-maker who will participate in the study
* Patient cognitively able to participate

Exclusion Criteria:

* Patient or their substitute decision-maker does not speak English
* Patient unable to identify a substitute decision-maker who will consent to participation
* Patient does not consent to participation

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 61 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Advance care planning engagement of substitute decision-maker | 8 to 12 weeks (6 weeks for patients from cancer centre)
  A survey of the substitute decision-maker's engagement in advance care planning

SECONDARY OUTCOMES:
Advance care planning engagement of patient | 8 to 12 weeks (6 weeks for patients from cancer centre)
  A survey of the patient's engagement in advance care planning
Substitute decision-maker self-efficacy survey | 8 to 12 weeks (6 weeks for patients from cancer centre)
  A survey of the substitute decision-maker's confidence to make future decisions
Decisional conflict | immediately after intervention
  A modified short decisional conflict survey
Satisfaction with intervention | immediately after intervention
  A satisfaction and endorsement survey on the process of the educational intervention

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Howard, PhD, Principal Investigator — McMaster University
Locations (7):
- Canada (7):
  - Dundas Family Health Team, Dundas, Ontario
  - Michael West Doctor Office, Dundas, Ontario
  - Burlington Family Health Team, Hamilton, Ontario
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - McMaster Family Health Team, Hamilton, Ontario
  - McMaster University Medical Centre, Hamilton, Ontario
  - Juravinski Cancer Centre Pain and Symptom Management Team, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] De Vleminck A, Houttekier D, Pardon K, Deschepper R, Van Audenhove C, Vander Stichele R, Deliens L. Barriers and facilitators for general practitioners to engage in advance care planning: a systematic review. Scand J Prim Health Care. 2013 Dec;31(4):215-26. doi: 10.3109/02813432.2013.854590. PMID 24299046
- [Result] Teixeira AA, Hanvey L, Tayler C, Barwich D, Baxter S, Heyland DK; Canadian Researchers at End of Life Network (CARENET). What do Canadians think of advanced care planning? Findings from an online opinion poll. BMJ Support Palliat Care. 2015 Mar;5(1):40-7. doi: 10.1136/bmjspcare-2013-000473. Epub 2013 Oct 4. PMID 24644188
- [Result] Howard M, Bernard C, Tan A, Slaven M, Klein D, Heyland DK. Advance care planning: Let's start sooner. Can Fam Physician. 2015 Aug;61(8):663-5. No abstract available. PMID 26273075
- [Result] Rhee JJ, Zwar NA, Kemp LA. Advance care planning and interpersonal relationships: a two-way street. Fam Pract. 2013 Apr;30(2):219-26. doi: 10.1093/fampra/cms063. Epub 2012 Oct 1. PMID 23028000
- [Result] Robinson C, Kolesar S, Boyko M, Berkowitz J, Calam B, Collins M. Awareness of do-not-resuscitate orders: what do patients know and want? Can Fam Physician. 2012 Apr;58(4):e229-33. PMID 22611610
- [Result] Sudore RL, Lum HD, You JJ, Hanson LC, Meier DE, Pantilat SZ, Matlock DD, Rietjens JAC, Korfage IJ, Ritchie CS, Kutner JS, Teno JM, Thomas J, McMahan RD, Heyland DK. Defining Advance Care Planning for Adults: A Consensus Definition From a Multidisciplinary Delphi Panel. J Pain Symptom Manage. 2017 May;53(5):821-832.e1. doi: 10.1016/j.jpainsymman.2016.12.331. Epub 2017 Jan 3. PMID 28062339
- [Result] Houben CHM, Spruit MA, Groenen MTJ, Wouters EFM, Janssen DJA. Efficacy of advance care planning: a systematic review and meta-analysis. J Am Med Dir Assoc. 2014 Jul;15(7):477-489. doi: 10.1016/j.jamda.2014.01.008. Epub 2014 Mar 2. PMID 24598477
- [Result] Teno JM, Fisher ES, Hamel MB, Coppola K, Dawson NV. Medical care inconsistent with patients' treatment goals: association with 1-year Medicare resource use and survival. J Am Geriatr Soc. 2002 Mar;50(3):496-500. doi: 10.1046/j.1532-5415.2002.50116.x. PMID 11943046
- [Result] Detering KM, Hancock AD, Reade MC, Silvester W. The impact of advance care planning on end of life care in elderly patients: randomised controlled trial. BMJ. 2010 Mar 23;340:c1345. doi: 10.1136/bmj.c1345. PMID 20332506
- [Result] Hammes BJ, Rooney BL. Death and end-of-life planning in one midwestern community. Arch Intern Med. 1998 Feb 23;158(4):383-90. doi: 10.1001/archinte.158.4.383. PMID 9487236
- [Result] Silveira MJ, Kim SY, Langa KM. Advance directives and outcomes of surrogate decision making before death. N Engl J Med. 2010 Apr 1;362(13):1211-8. doi: 10.1056/NEJMsa0907901. PMID 20357283
- [Result] Raymont V, Bingley W, Buchanan A, David AS, Hayward P, Wessely S, Hotopf M. Prevalence of mental incapacity in medical inpatients and associated risk factors: cross-sectional study. Lancet. 2004 Oct 16-22;364(9443):1421-7. doi: 10.1016/S0140-6736(04)17224-3. PMID 15488217
- [Result] Fried TR, Redding CA, Robbins ML, O'Leary JR, Iannone L. Agreement between older persons and their surrogate decision-makers regarding participation in advance care planning. J Am Geriatr Soc. 2011 Jun;59(6):1105-9. doi: 10.1111/j.1532-5415.2011.03412.x. Epub 2011 Jun 7. PMID 21649619
- [Result] Heyland DK, Ilan R, Jiang X, You JJ, Dodek P. The prevalence of medical error related to end-of-life communication in Canadian hospitals: results of a multicentre observational study. BMJ Qual Saf. 2016 Sep;25(9):671-9. doi: 10.1136/bmjqs-2015-004567. Epub 2015 Nov 9. PMID 26554026
- [Result] You JJ, Dodek P, Lamontagne F, Downar J, Sinuff T, Jiang X, Day AG, Heyland DK; ACCEPT Study Team and the Canadian Researchers at the End of Life Network (CARENET). What really matters in end-of-life discussions? Perspectives of patients in hospital with serious illness and their families. CMAJ. 2014 Dec 9;186(18):E679-87. doi: 10.1503/cmaj.140673. Epub 2014 Nov 3. PMID 25367427
- [Result] Heyland DK, Barwich D, Pichora D, Dodek P, Lamontagne F, You JJ, Tayler C, Porterfield P, Sinuff T, Simon J; ACCEPT (Advance Care Planning Evaluation in Elderly Patients) Study Team; Canadian Researchers at the End of Life Network (CARENET). Failure to engage hospitalized elderly patients and their families in advance care planning. JAMA Intern Med. 2013 May 13;173(9):778-87. doi: 10.1001/jamainternmed.2013.180. PMID 23545563
- [Result] Cook D, Rocker G, Marshall J, Sjokvist P, Dodek P, Griffith L, Freitag A, Varon J, Bradley C, Levy M, Finfer S, Hamielec C, McMullin J, Weaver B, Walter S, Guyatt G; Level of Care Study Investigators and the Canadian Critical Care Trials Group. Withdrawal of mechanical ventilation in anticipation of death in the intensive care unit. N Engl J Med. 2003 Sep 18;349(12):1123-32. doi: 10.1056/NEJMoa030083. PMID 13679526
- [Result] Gruneir A, Mor V, Weitzen S, Truchil R, Teno J, Roy J. Where people die: a multilevel approach to understanding influences on site of death in America. Med Care Res Rev. 2007 Aug;64(4):351-78. doi: 10.1177/1077558707301810. PMID 17684107
- [Result] Heyland DK, Lavery JV, Tranmer JE, Shortt SE, Taylor SJ. Dying in Canada: is it an institutionalized, technologically supported experience? J Palliat Care. 2000 Oct;16 Suppl:S10-6. PMID 11075528
- [Result] Ehlenbach WJ, Barnato AE, Curtis JR, Kreuter W, Koepsell TD, Deyo RA, Stapleton RD. Epidemiologic study of in-hospital cardiopulmonary resuscitation in the elderly. N Engl J Med. 2009 Jul 2;361(1):22-31. doi: 10.1056/NEJMoa0810245. PMID 19571280
- [Derived] Howard M, Elston D, Borhan S, Hafid A, Arora N, Forbes R, Bernard C, Heyland DK. Randomised trial of a serious illness decision aid (Plan Well Guide) for patients and their substitute decision-makers to improve engagement in advance care planning. BMJ Support Palliat Care. 2022 Mar;12(1):99-106. doi: 10.1136/bmjspcare-2021-003040. Epub 2021 Jun 30. PMID 34193434
- [Derived] Howard M, Slaven M, Bernard C, Borhan S, Elston D, Arora N, Tan A, Heyland DK. Decision support intervention (Plan Well Guide) for patients and their substitute decision-makers to improve engagement in advance care planning: protocol for a randomised trial. BMJ Open. 2019 Sep 20;9(9):e027897. doi: 10.1136/bmjopen-2018-027897. PMID 31542737
- See also: Metzger M, Song M-K, Ward S, Chang PP-Y, Hanson LC, Lin F-C. A randomized controlled pilot trial to improve advance care planning for LVAD patients and their surrogates. Hear Lung J Acute Crit Care. 2016 May;45(3):186-92 — http://www.ncbi.nlm.nih.gov/pubmed/26948697
- See also: Johnston SC, Pfeifer MP, McNutt R. The discussion about advance directives. Patient and physician opinions regarding when and how it should be conducted. End of Life Study Group. Arch Intern Med. 1995 May 22;155(10):1025-30 — http://www.ncbi.nlm.nih.gov/pubmed/7748044
- See also: Rhee JJ, Zwar NA, Kemp LA. Advance care planning and interpersonal relationships: a two-way street. Fam Pract. 2013 Apr 1;30(2):219-26 — http://www.ncbi.nlm.nih.gov/pubmed/23028000